CLINICAL TRIAL: NCT01595672
Title: Early High-volume Continuous Veno-venous Hemofiltration for Patients With Severe Acute Pancreatitis: Single-center, Randomized, Controlled Trial
Brief Title: Early High-volume Continuous Veno-venous Hemofiltration for Patients With Severe Acute Pancreatitis
Acronym: EHVCVVHSAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Qingchuan Zhao, Clinical Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAP-CVVH-XHDD-002; 81170432 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2012-05-04; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Acute Pancreatitis
Keywords: severe acute pancreatitis; organ failure; multiple organ dysfunction syndrome; systemic complications; continuous veno-venous hemofiltration; blood purification; continuous renal replacement therapy
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EHVCVVH group (Active Comparator): Patients receive conventional treatments recommended by guidelines with adjunctive early high-volume continuous veno-venous hemofiltration (EHVCVVH).
  Interventions: Device: AN69 hemofilter
- Control group (Active Comparator): Patients receive conventional treatments recommended by guidelines only.
  Interventions: Other: conventional treatments

INTERVENTIONS:
Device: AN69 hemofilter — An AN69 hemofilter (1.6 m2 surface area, 35-KD limit; Baxter Healthcare Corp. Deerfield, IL, USA) will be used for EHCVVH.
  Other Names: high-volume hemofiltration
  Arms: EHVCVVH group
Other: conventional treatments — Patients receive conventional treatments recommended by guidelines only.
  Other Names: standard treatments
  Arms: Control group

SUMMARY:
The purpose of this study is to determine the effect and safety of early high-volume continuous veno-venous hemofiltration for patients with severe acute pancreatitis.

DETAILED DESCRIPTION:
The investigators anticipated that early high-volume continuous veno-venous hemofiltration (EHVCVVH) would result in a decrease of the composite of persistent organ failure or death by eliminating inflammatory mediators in blood. This study is designed to evaluate the impact of EHVCVVH on patients with severe acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of severe acute pancreatitis
* written informed consent
* Time from onset of abdominal pain to admission ≤ 72 hours
* SIRS score ≥ 2

Exclusion Criteria:

* confirmed infection
* pregnancy
* patients needing emergency operation for abdominal compartment syndrome
* chronic renal diseases needing blood purification
* previous exploratory laparotomy for acute abdomen and diagnosis of pancreatitis during laparotomy
* acute flare-up of chronic pancreatitis
* malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
persistent organ failure or death | 1 months
  persistent organ failure: organ failure ≥ 48 hours

SECONDARY OUTCOMES:
death | 1 months
persistent organ failure | 1 months
infectious complications | 1 months
  infected necrosis,bacteraemia and pneumonia respectively
input fluid volume within first 3 days after admission | 3 days
  crystalloid fluids and colloid fluids respectively
Physiological Parameters 1 day, 2 days, and 3 days after randomization | 3 days
  Physiological Parameters: APACHE-II score,SOFA score,Body temperature,PaO2/FiO2,BE,PLT,Cr,serum Ca,WBC and Urine volume
The concentration of inflammatory mediators in serum 0 hour,2 hours,6 hours and 12 hours after early high-volume continuous veno-venous hemofiltration | 12 hours
  inflammatory mediators: tumor necrosis factor-α, IL-1, IL-2, IL-4, IL-6, and IL-8, IL-10, IL-13, IL-15, Angiopoietin-2, trypsin, resistin and visfatin
total number of surgical interventions | 2 months
  for any purpose
ICU stay | 2 months
total costs in hospital | 3 months
output fluid volume in the first, second, third day after admission | 3 days
  output: urine volume,ultrafiltration liquids,gastric drainage and defecation
persistent multiple organ dysfunction syndrome | 1 months
  multiple organ dysfunction syndrome (two or more organs or occurrence of two or more systemic complications at the same time) ≥ 48 hours
new-onset organ failure | 1 months
  not present at any time in the 24 hours before randomization
new-onset multiple organ dysfunction syndrome | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Qingchuan, PhD & MD, Principal Investigator — the First Affiliated Hospital of Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China